CLINICAL TRIAL: NCT01122238
Title: Identifying Optimal, Translatable Smoking Cessation Intervention Components
Brief Title: Identifying Treatments to Motivate Smokers to Quit
Acronym: Motivation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of Illinois at Chicago (Other); Dean Health System (Other); Mercy Health System (Network); Wake Forest University Health Sciences (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: H-2009-0203; 9P50CA143188 (NIH)
Record Dates: First submitted 2010-05-07; First posted 2010-05-13 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-11

CONDITIONS: Smoking; Smoking Cessation; Motivation; Nicotine Dependence
Keywords: Smoking; Smoking Cessation; Motivation; Nicotine Dependence
MeSH Terms: conditions — Smoking; Smoking Cessation; Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices; Nicotine Chewing Gum; Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (16):
- 1, Nicotine Patch, Nicotine Gum, Reduction, MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? Nicotine Patch, Nicotine Gum, Smoking Reduction Counseling, and Motivational Interviewing (MI)
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Smoking Reduction; Drug: Nicotine Patch + Nicotine Gum
- 2, Nicotine Patch, Nicotine Gum, Reduction, No MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? Nicotine Patch, Nicotine Gum, Smoking Reduction Counseling, and No Motivational Interviewing (MI)
  Interventions: Behavioral: Motivational Interviewing; Drug: Nicotine Patch + Nicotine Gum
- 3, Nicotine Patch, Nicotine Gum, No Reduction, MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? Nicotine Patch, Nicotine Gum, No Smoking Reduction Counseling, and Motivational Interviewing (MI)
  Interventions: Behavioral: Smoking Reduction; Drug: Nicotine Patch + Nicotine Gum
- 4, Nicotine Patch, Nicotine Gum, No Reduction, No MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? Nicotine Patch, Nicotine Gum, No Smoking Reduction Counseling, and No Motivational Interviewing (MI)
  Interventions: Drug: Nicotine Patch + Nicotine Gum
- 5, Nicotine Patch, No Nicotine Gum, Reduction, MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? Nicotine Patch, No Nicotine Gum, Smoking Reduction Counseling, and Motivational Interviewing (MI)
  Interventions: Drug: Nicotine Patch; Behavioral: Motivational Interviewing; Behavioral: Smoking Reduction
- 6, Nicotine Patch, No Nicotine Gum, Reduction, No MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? Nicotine Patch, No Nicotine Gum, Smoking Reduction Counseling, and No Motivational Interviewing (MI)
  Interventions: Drug: Nicotine Patch; Behavioral: Motivational Interviewing
- 7, Nicotine Patch, No Nicotine Gum, No Reduction, MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? Nicotine Patch, No Nicotine Gum, No Smoking Reduction Counseling, and Motivational Interviewing (MI)
  Interventions: Drug: Nicotine Patch; Behavioral: Smoking Reduction
- 8, Nicotine Patch, No Nicotine Gum, No Reduction, No MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? Nicotine Patch, No Nicotine Gum, No Smoking Reduction Counseling, and No Motivational Interviewing (MI)
  Interventions: Drug: Nicotine Patch
- 9, No Nicotine Patch, Nicotine Gum, Reduction, MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? No Nicotine Patch, Nicotine Gum, Smoking Reduction Counseling, and Motivational Interviewing (MI)
  Interventions: Drug: Nicotine Gum; Behavioral: Motivational Interviewing; Behavioral: Smoking Reduction
- 10, No Nicotine Patch, Nicotine Gum, Reduction, No MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? No Nicotine Patch, Nicotine Gum, Smoking Reduction Counseling, and No Motivational Interviewing (MI)
  Interventions: Drug: Nicotine Gum; Behavioral: Motivational Interviewing
- 11, No Nicotine Patch, Nicotine Gum, No Reduction, MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? No Nicotine Patch, Nicotine Gum, No Smoking Reduction Counseling, and Motivational Interviewing (MI)
  Interventions: Drug: Nicotine Gum; Behavioral: Smoking Reduction
- 12, No Nicotine Patch, Nicotine Gum, No Reduction, No MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? No Nicotine Patch, Nicotine Gum, No Smoking Reduction Counseling, and No Motivational Interviewing (MI)
  Interventions: Drug: Nicotine Gum
- 13, No Nicotine Patch, No Nicotine Gum, Reduction, MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? No Nicotine Patch, No Nicotine Gum, Smoking Reduction Counseling, and Motivational Interviewing (MI)
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Smoking Reduction
- 14, No Nicotine Patch, No Nicotine Gum, Reduction, No MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? No Nicotine Patch, No Nicotine Gum, Smoking Reduction Counseling, and No Motivational Interviewing (MI)
  Interventions: Behavioral: Motivational Interviewing
- 15, No Nicotine Patch, No Nicotine Gum, No Reduction, MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? No Nicotine Patch, No Nicotine Gum, No Smoking Reduction Counseling, and Motivational Interviewing (MI)
  Interventions: Behavioral: Smoking Reduction
- 16, No Nicotine Patch, No Nicotine Gum, No Reduction, No MI (Experimental): This arm of the project will address the following question:
  How effective is the following intervention? No Nicotine Patch, No Nicotine Gum, No Smoking Reduction Counseling, and No Motivational Interviewing (MI)
  Interventions: Other: No Intervention

INTERVENTIONS:
Drug: Nicotine Patch — If randomized to only the Nicotine Patch condition (and not the Nicotine Gum):
  Participants randomized to this condition will receive a 6-week supply of 14 mg patches at the initial visit. Participant will be instructed to use one patch daily for 6 weeks.
  Arms: 5, Nicotine Patch, No Nicotine Gum, Reduction, MI; 6, Nicotine Patch, No Nicotine Gum, Reduction, No MI; 7, Nicotine Patch, No Nicotine Gum, No Reduction, MI; 8, Nicotine Patch, No Nicotine Gum, No Reduction, No MI
Drug: Nicotine Gum — If randomized to only the Nicotine Gum condition (and not the Nicotine Patch):
  Participants randomized to this condition will receive a 6-week supply of 2 mg gum at the initial visit. Participants will be instructed to use 10 pieces of gum daily for 6 weeks.
  Arms: 10, No Nicotine Patch, Nicotine Gum, Reduction, No MI; 11, No Nicotine Patch, Nicotine Gum, No Reduction, MI; 12, No Nicotine Patch, Nicotine Gum, No Reduction, No MI; 9, No Nicotine Patch, Nicotine Gum, Reduction, MI
Behavioral: Motivational Interviewing — Participants randomized to this condition will receive an initial MI counseling session during the in-person clinic visit followed by three counseling phone calls over the 6-week intervention period (a total of four intervention contacts). The phone counseling sessions will occur during weeks 2, 4, and 6. Case managers will engage the participant in a series of motivation building exercises such as reviewing feelings and thoughts about the pros and cons of quitting and smoking, reinforcing the positives of quitting, helping to dispel myths and concerns about the negatives of quitting, and posing questions about the "good" aspects of smoking.
  Arms: 1, Nicotine Patch, Nicotine Gum, Reduction, MI; 10, No Nicotine Patch, Nicotine Gum, Reduction, No MI; 13, No Nicotine Patch, No Nicotine Gum, Reduction, MI; 14, No Nicotine Patch, No Nicotine Gum, Reduction, No MI; 2, Nicotine Patch, Nicotine Gum, Reduction, No MI; 5, Nicotine Patch, No Nicotine Gum, Reduction, MI; 6, Nicotine Patch, No Nicotine Gum, Reduction, No MI; 9, No Nicotine Patch, Nicotine Gum, Reduction, MI
Behavioral: Smoking Reduction — Participants randomized to Smoking Reduction will receive an initial counseling session during the in-person visit followed by 6 weekly phone counseling sessions over the 6-week intervention period. During the initial session, participants will be told that the goal is to reduce cigarette consumption by 50% over the course of the intervention (approximately 10% reduction per week). During the initial meeting and subsequent counseling calls, case managers will work with participants to problem-solve strategies for reduction (e.g., increasing time between cigarettes, delaying smoking, or eliminating smoking in specific situations). Participants will be asked to record information in a provided smoking log to help keep track of daily smoking patterns and as a feedback mechanism for identifying successes and challenges.
  Arms: 1, Nicotine Patch, Nicotine Gum, Reduction, MI; 11, No Nicotine Patch, Nicotine Gum, No Reduction, MI; 13, No Nicotine Patch, No Nicotine Gum, Reduction, MI; 15, No Nicotine Patch, No Nicotine Gum, No Reduction, MI; 3, Nicotine Patch, Nicotine Gum, No Reduction, MI; 5, Nicotine Patch, No Nicotine Gum, Reduction, MI; 7, Nicotine Patch, No Nicotine Gum, No Reduction, MI; 9, No Nicotine Patch, Nicotine Gum, Reduction, MI
Other: No Intervention — No Intervention
  Arms: 16, No Nicotine Patch, No Nicotine Gum, No Reduction, No MI
Drug: Nicotine Patch + Nicotine Gum — If randomized to both the Nicotine Patch and the Nicotine Gum conditions:
  Participants randomized to this condition will receive a 6-week supply of 14 mg patches and a 6-week supply of 2 mg gum at the initial visit. Participant will be instructed to use one patch daily and to use 10 pieces of gum daily for 6 weeks.
  Arms: 1, Nicotine Patch, Nicotine Gum, Reduction, MI; 2, Nicotine Patch, Nicotine Gum, Reduction, No MI; 3, Nicotine Patch, Nicotine Gum, No Reduction, MI; 4, Nicotine Patch, Nicotine Gum, No Reduction, No MI

SUMMARY:
At any given point in time, most smokers are not interested in making a serious quit attempt. Data suggest that 30% of smokers have no plans to quit, 30% plan to quit at some future date, 30% plan to quit in the next 6 months, and about 10% plan to quit in the next month. While ~40% of smokers make a quit attempt each year, only about 4-6% of those achieve long-term success. This means that of the more than 60 million Americans who smoke, only 1 million are able to quit each year. If we could double the number of quit attempts and maintain comparable success rates, we could double the number of individuals who will benefit from living smoke free lives. These observations underscore the need to develop interventions that increase smokers' motivation or willingness to make quit attempts, and that also increase the rate of success among those who attempt to quit. The overall goal of this proposed experiment is to identify effective interventions aimed at increasing motivation for smoking cessation, increasing quit attempts, and increasing rates of cessation success. Interventions that will be tested include: use of nicotine gum, use of nicotine patches, motivational interviewing, and smoking reduction counseling. At minimum, all participants will complete surveys about their smoking behavior that might increase their motivation to eventually quitting smoking.

DETAILED DESCRIPTION:
This study used efficient research methods to screen four intervention components (Nicotine Patch, Nicotine Gum, Motivational Interviewing, Behavioral Reduction Counseling) that were designed to reduce smoking heaviness, enhance quitting success, and be easily translated into healthcare settings. These components were evaluated amongst smokers recruited in primary care who were unwilling to make a quit attempt, but who were willing to reduce their smoking. The main objective was to identify promising Motivation phase components for inclusion in a comprehensive chronic care smoking treatment.

Recruitment and Enrollment:

Participants were recruited from 11 primary care clinics in southern Wisconsin using existing rooming staff (i.e., medical assistants) who were prompted by electronic health record technology. During clinic visits, identified smokers were invited to participate in a research program to help them reduce their smoking. Interested patients were electronically referred to the research office. Research staff contacted interested patients and assessed eligibility. Eligible patients were invited to return to their primary care clinic to learn about the study, provide written informed consent, be randomized, and complete initial assessments. A database created a schedule of intervention and assessment contacts, which guided treatment delivery by case managers. The case managers in this study were bachelor's level research staff.

There was an initial 6-week Motivation phase treatment period, and participants could choose to extend the treatment for another 6 weeks (so Motivation phase treatment lasted either 6 or 12 weeks). Participants who chose to extend the treatment continued to receive the same components to which they were originally, randomly assigned. In addition, participants could elect to receive Cessation phase treatment at any point throughout the 6-month study period. Cessation phase treatment was identical for all participants and consisted of 8 weeks of nicotine patch + nicotine gum, and two brief phone counseling sessions.

Study Design:

This 2x2x2x2 factorial experiment had four factors each comprising an active (ON) condition and control (OFF) condition: 1) Nicotine Patch; 2) Nicotine Gum; 3) Motivational Interviewing; and 4) Behavioral Reduction Counseling, yielding 16 unique combinations of experimental conditions. Subjects were randomly assigned to one of the 16 experimental conditions, stratifying by gender. All treatment components were designed to be compatible with one another, and to be delivered with fidelity across all treatment combinations.

Experimental Factors:

Nicotine Patch vs. No Patch. Participants in the ON (active) condition were instructed to use 14-mg patches daily for the 6-week intervention period.

Nicotine Gum vs. No Gum. Participants in the ON condition were instructed to use 2-mg nicotine gum for the 6-week intervention period (≥9/day, 1 piece/1-2 hours) in place of smoking.

Motivational Interviewing (MI) vs. No MI. Participants in the ON condition received an initial 20-minute in-person counseling session followed by three 20-minute counseling calls over the 6-week intervention period. As per Miller and Rollnick (50, 51), the counseling sessions included motivation-building exercises to reinforce intrinsic motivation and to help participants overcome ambivalence about quitting.

Behavioral Reduction (BR) vs. No BR. Participants in the ON condition received an initial 20-minute in-person counseling session followed by 6 weekly 20-minute counseling calls. During these sessions, participants set smoking reduction goals and developed reduction strategies (e.g., delaying smoking, eliminating smoking in specific situations). Participants were also instructed to record daily smoking, which case managers used to identify successes and challenges.

Assessments:

Participants completed baseline assessments of vital signs, demographics, and smoking history and dependence (e.g., the Fagerström Test for Nicotine Dependence). During study visits, adverse events, medication adherence, and smoking in the past week were assessed. The last was used to determine the primary outcome of cigarettes smoked per day (CPD) at 12 and 26 weeks, as well as 7-day point-prevalence abstinence (no smoking for the past 7 days) at 26 weeks post study entry. Smoking heaviness reflects both smoking reduction and abstinence, and thus captures the net impact of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Report smoking at least 5 cigarettes per day for the previous 6 months;
* Able to read and write English;
* Available to take one phone call per week;
* Not currently interested in quitting smoking (defined as would not like to try to quit in the next 30 days),
* Plans to remain in the intervention catchment area for at least 12 months
* All women of childbearing potential will be required to agree to use an acceptable method of birth control to prevent pregnancy during the study.

Exclusion Criteria:

* Currently taking bupropion, Wellbutrin, chantix or varenicline (current use of NRT is not exclusionary if the participant agrees to use only study medication for the duration of the study);
* Study candidate is a pregnant, trying to get pregnant, or nursing;
* A history of psychosis or bipolar disorder
* A history of skin or allergic reactions while using a nicotine patch.
* Study candidate reports having a heart attack, stroke, or abnormal electrocardiogram within the past 4 weeks.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2010-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C. Fiore, MD, MPH, MBA, Study Chair — University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health; Jessica Cook, PhD, Study Director — University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health; Robin Mermelstein, PhD, Principal Investigator — Institute for Health Research and Policy, University of Illinois at Chicago
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995
- See also: University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health — http://www.ctri.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1, Nicotine Patch, Nicotine Gum, Reduction, MI | 2, Nicotine Patch, Nicotine Gum, Reduction, No MI | 3, Nicotine Patch, Nicotine Gum, No Reduction, MI | 4, Nicotine Patch, Nicotine Gum, No Reduction, No MI | 5, Nicotine Patch, No Nicotine Gum, Reduction, MI | 6, Nicotine Patch, No Nicotine Gum, Reduction, No MI | 7, Nicotine Patch, No Nicotine Gum, No Reduction, MI | 8, Nicotine Patch, No Nicotine Gum, No Reduction, No MI | 9, No Nicotine Patch, Nicotine Gum, Reduction, MI | 10, No Nicotine Patch, Nicotine Gum, Reduction, No MI | 11, No Nicotine Patch, Nicotine Gum, No Reduction, MI | 12, No Nicotine Patch, Nicotine Gum, No Reduction, No MI | 13, No Nicotine Patch, No Nicotine Gum, Reduction, MI | 14, No Nicotine Patch, No Nicotine Gum, Reduction, No MI | 15, No Nicotine Patch, No Nicotine Gum, No Reduction, MI | 16, No Nicotine Patch, No Nicotine Gum, No Reduction, No MI
Started | 30 | 37 | 33 | 33 | 33 | 32 | 35 | 32 | 32 | 34 | 32 | 33 | 30 | 32 | 28 | 31
Completed | 28 | 36 | 28 | 33 | 33 | 31 | 34 | 32 | 31 | 33 | 32 | 31 | 28 | 31 | 28 | 31
Not Completed | 2 | 1 | 5 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Adult smokers who consented to enroll in the treatment study.
Groups:
- Total: Total of all reporting groups
Arm/Group | 1, Nicotine Patch, Nicotine Gum, Reduction, MI | 2, Nicotine Patch, Nicotine Gum, Reduction, No MI | 3, Nicotine Patch, Nicotine Gum, No Reduction, MI | 4, Nicotine Patch, Nicotine Gum, No Reduction, No MI | 5, Nicotine Patch, No Nicotine Gum, Reduction, MI | 6, Nicotine Patch, No Nicotine Gum, Reduction, No MI | 7, Nicotine Patch, No Nicotine Gum, No Reduction, MI | 8, Nicotine Patch, No Nicotine Gum, No Reduction, No MI | 9, No Nicotine Patch, Nicotine Gum, Reduction, MI | 10, No Nicotine Patch, Nicotine Gum, Reduction, No MI | 11, No Nicotine Patch, Nicotine Gum, No Reduction, MI | 12, No Nicotine Patch, Nicotine Gum, No Reduction, No MI | 13, No Nicotine Patch, No Nicotine Gum, Reduction, MI | 14, No Nicotine Patch, No Nicotine Gum, Reduction, No MI | 15, No Nicotine Patch, No Nicotine Gum, No Reduction, MI | 16, No Nicotine Patch, No Nicotine Gum, No Reduction, No MI | Total
Number analyzed (Participants) | 30 | 37 | 33 | 33 | 33 | 32 | 35 | 32 | 32 | 34 | 32 | 33 | 30 | 32 | 28 | 31 | 517
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 6
  Between 18 and 65 years | 29 | 34 | 27 | 26 | 32 | 30 | 30 | 28 | 29 | 30 | 26 | 31 | 25 | 27 | 22 | 26 | 452
  >=65 years | 1 | 3 | 5 | 7 | 1 | 2 | 4 | 3 | 3 | 4 | 4 | 2 | 5 | 4 | 6 | 5 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.37 (13.28) | 46.00 (14.05) | 49.18 (14.89) | 48.91 (13.22) | 47.00 (14.03) | 48.47 (14.50) | 44.89 (14.57) | 47.91 (14.19) | 41.63 (15.40) | 49.53 (13.77) | 45.41 (14.89) | 47.30 (13.90) | 46.87 (14.71) | 47.06 (14.98) | 51.93 (12.82) | 46.84 (15.18) | 47.05 (14.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 20 | 21 | 21 | 19 | 23 | 21 | 20 | 21 | 21 | 22 | 18 | 21 | 18 | 19 | 328
  Male | 11 | 13 | 13 | 12 | 12 | 13 | 12 | 11 | 12 | 13 | 11 | 11 | 12 | 11 | 10 | 12 | 189
Region of Enrollment [Number; unit: participants]
  United States | 30 | 37 | 33 | 33 | 33 | 32 | 35 | 32 | 32 | 34 | 32 | 33 | 30 | 32 | 28 | 31 | 517

OUTCOME MEASURES:

1. Secondary Outcome: Average Number of Cigarettes Per Day in the Past Week.
Time Frame: Assessed at baseline and week 26.
Population: Adult smokers not yet motivated to quit smoking. The project design measured change in the smoking patterns of these individuals.
Measure: Mean (Standard Deviation); unit: Change in cigarettes per day
Groups:
- Nicotine Patch: All participants in this group received Nicotine Patch; the group includes participants who received combinations of the other three study interventions (Nicotine Gum or No Nicotine Gum; Motivational Interviewing or No Motivational Interviewing); Smoking Reduction or No Smoking Reduction). The Nicotine Patch group consists of 265 participants (approximately half of the total study sample) and will be compared to a corresponding No Nicotine Patch group consisting of 252 participants (approximately half of the total study sample) in a main effect (Nicotine Patch versus No Nicotine Patch) statistical comparison.
- No Nicotine Patch: All participants in this group received No Nicotine Patch; the group includes participants who received combinations of the other three study interventions (Nicotine Gum or No Nicotine Gum; Motivational Interviewing or No Motivational Interviewing); Smoking Reduction or No Smoking Reduction). The No Nicotine Patch group consists of 252 participants (approximately half of the total study sample) and will be compared to a corresponding Nicotine Patch group consisting of 265 participants (approximately half of the total study sample) in a main effect (Nicotine Patch versus No Nicotine Patch) statistical comparison.
- Nicotine Gum: All participants in this group received Nicotine Gum; the group includes participants who received combinations of the other three study interventions (Nicotine Patch or No Nicotine Patch; Motivational Interviewing or No Motivational Interviewing); Smoking Reduction or No Smoking Reduction). The Nicotine Gum group consists of 264 participants (approximately half of the total study sample) and will be compared to a corresponding No Nicotine Gum group consisting of 253 participants (approximately half of the total study sample) in a main effect (Nicotine Gum versus No Nicotine Gum) statistical comparison.
- No Nicotine Gum: All participants in this group received No Nicotine Gum; the group includes participants who received combinations of the other three study interventions (Nicotine Patch or No Nicotine Patch; Motivational Interviewing or No Motivational Interviewing); Smoking Reduction or No Smoking Reduction). The No Nicotine Gum group consists of 253 participants (approximately half of the total study sample) and will be compared to a corresponding Nicotine Gum group consisting of 264 participants (approximately half of the total study sample) in a main effect (Nicotine Gum versus No Nicotine Gum) statistical comparison.
- Smoking Reduction: All participants in this group received Smoking Reduction counseling; the group includes participants who received combinations of the other three study interventions (Nicotine Patch or No Nicotine Patch; Nicotine Gum or No Nicotine Gum; Motivational Interviewing or No Motivational Interviewing). The Smoking Reduction group consists of 260 participants (approximately half of the total study sample) and will be compared to a corresponding No Smoking Reduction group consisting of 257 participants (approximately half of the total study sample) in a main effect (Smoking Reduction versus No Smoking Reduction) statistical comparison.
- No Smoking Reduction: All participants in this group received No Smoking Reduction counseling; the group includes participants who received combinations of the other three study interventions (Nicotine Patch or No Nicotine Patch; Nicotine Gum or No Nicotine Gum; Motivational Interviewing or No Motivational Interviewing). The No Smoking Reduction group consists of 257 participants (approximately half of the total study sample) and will be compared to a corresponding Smoking Reduction group consisting of 260 participants (approximately half of the total study sample) in a main effect (Smoking Reduction versus No Smoking Reduction) statistical comparison.
- Motivational Interviewing: All participants in this group received Motivational Interviewing counseling; the group includes participants who received combinations of the other three study interventions (Nicotine Patch or No Nicotine Patch; Nicotine Gum or No Nicotine Gum; Smoking Reduction or No Smoking Reduction). The Motivational Interviewing group consists of 253 participants (approximately half of the total study sample) and will be compared to a corresponding No Motivational Interviewing group consisting of 264 participants (approximately half of the total study sample) in a main effect (Motivational Interviewing versus No Motivational Interviewing) statistical comparison.
- No Motivational Interviewing: All participants in this group received No Motivational Interviewing counseling; the group includes participants who received combinations of the other three study interventions (Nicotine Patch or No Nicotine Patch; Nicotine Gum or No Nicotine Gum; Smoking Reduction or No Smoking Reduction). The No Motivational Interviewing group consists of 264 participants (approximately half of the total study sample) and will be compared to a corresponding Motivational Interviewing group consisting of 253 participants (approximately half of the total study sample) in a main effect (Motivational Interviewing versus No Motivational Interviewing) statistical comparison.
Arm/Group | Nicotine Patch | No Nicotine Patch | Nicotine Gum | No Nicotine Gum | Smoking Reduction | No Smoking Reduction | Motivational Interviewing | No Motivational Interviewing
Number analyzed (Participants) | 265 | 252 | 264 | 253 | 260 | 257 | 253 | 264
Change in cigarettes per day | .117 (6.688) | -.123 (6.540) | .179 (6.402) | -.187 (6.830) | -.158 (6.568) | .160 (6.663) | .371 (6.597) | -.353 (6.617)
Statistical Analysis 1: Comparison: Nicotine Patch vs No Nicotine Patch; The ANCOVA model included intervention main effects and intervention interactions plus baseline cigarettes per day, education, race, and time to first daily cigarette as covariates. Intervention main effects included Nicotine Patch vs. No Nicotine Patch; Nicotine Gum vs. No Nicotine Gum; Smoking Reduction vs. No Smoking Reduction; and Motivational Interviewing vs. No Motivational Interviewing; Test type: Superiority or Other; p = .665, ANCOVA; The mean values tested and reported consist of residualized change scores from the ANCOVA
Statistical Analysis 2: Comparison: Nicotine Gum vs No Nicotine Gum; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .562, ANCOVA; The mean values tested and reported consist of residualized change scores from the ANCOVA
Statistical Analysis 3: Comparison: Smoking Reduction vs No Smoking Reduction; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .536, ANCOVA; The mean values tested and reported consist of residualized change scores from the ANCOVA
Statistical Analysis 4: Comparison: Motivational Interviewing vs No Motivational Interviewing; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = .206, ANCOVA; The mean values tested and reported consist of residualized change scores from the ANCOVA

2. Primary Outcome: Percent Change in Cigarettes Smoked Per Day (CPD)
Description: Percent Change in Cigarettes Smoked Per Day (CPD) is computed as the percent change in self-reported cigarettes smoked per day at the assessment endpoint relative to baseline CPD; this outcome will be analyzed in a linear regression analysis model.
  Note: This Percent change in Cigarettes Smoked Per Day (CPD) primary outcome replaces "average number of cigarettes per day in the past week" (now designated as a secondary outcome) because the percent change metric allows better comparison with prior research in this area and the results for both outcomes are highly similar.
Time Frame: Assessed at week 26 relative to baseline CPD.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change in cigarettes per day
Arm/Group | Nicotine Patch | No Nicotine Patch | Nicotine Gum | No Nicotine Gum | Smoking Reduction | No Smoking Reduction | Motivational Interviewing | No Motivational Interviewing
Number analyzed (Participants) | 265 | 252 | 264 | 253 | 260 | 257 | 253 | 264
Percent Change in cigarettes per day | 38.7 (36.2) | 38.9 (37.1) | 37.4 (36.2) | 40.2 (36.9) | 38.6 (36.3) | 38.9 (36.9) | 37.2 (35.6) | 40.2 (37.5)
Statistical Analysis 1: Comparison: Nicotine Patch vs No Nicotine Patch; The linear regression model effects consisted of four treatment main effects, six two-way treatment interactions, four three-way treatment interactions, and one four-way interaction. Only the results for the treatment main effects are being reported in ClinicalTrials.gov; Test type: Superiority or Other; p = .98, Regression, Linear; Standardized Regression Coefficient = -.00
Statistical Analysis 2: Comparison: Nicotine Gum vs No Nicotine Gum; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .40, Regression, Linear; Standardized Regression Coefficient = -.04
Statistical Analysis 3: Comparison: Smoking Reduction vs No Smoking Reduction; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .99, Regression, Linear; Standardized Regression Coefficient = -.00
Statistical Analysis 4: Comparison: Motivational Interviewing vs No Motivational Interviewing; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = .33, Regression, Linear; Standardized Regression Coefficient = -.04

ADVERSE EVENTS:
Time Frame: AEs were reported weekly for the 6 weeks study subjects were on medication.
Description: Data from ad Hoc AE reports and protocol prompted weekly AE assessments were combined. Only AEs where 5% or more of those from a study arm were reported and compared to other study arms.
Groups:
- Prequit Combined Nicotine Patch + Gum: Prequit Combined Nicotine Patch + Gum
  Participants randomized to this condition received a 6-week supply of 14 mg patches and a 6-week supply of 2 mg gum at the initial visit. Participant will be instructed to use one patch daily and to use 10 pieces of gum daily for 6 weeks.
- Prequit Nicotine Patch Only: Prequit Nicotine Patch Only
  Participants randomized to this condition received a 6-week supply of 14 mg patches at the initial visit. Participant will be instructed to use one patch daily for 6 weeks.
- Prequit Nicotine Gum Only: Prequit Nicotine Gum Only.
  Participants randomized to this condition received a 6-week supply of 2 mg gum at the initial visit. Participants will be instructed to use 10 pieces of gum daily for 6 weeks.
- No Medication: No Medication
  Participants randomized to this condition received no medication.
Arm/Group | Prequit Combined Nicotine Patch + Gum | Prequit Nicotine Patch Only | Prequit Nicotine Gum Only | No Medication
Serious Adverse Events (participants affected / at risk) | 2/133 | 1/132 | 3/131 | 2/121
Other Adverse Events (participants affected / at risk) | 71/133 | 67/132 | 33/131 | 0/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prequit Combined Nicotine Patch + Gum (N=133) | Prequit Nicotine Patch Only (N=132) | Prequit Nicotine Gum Only (N=131) | No Medication (N=121)
Cardiovascular (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) — specific Adverse Event Terms are unknown because adverse events were only collected with regard to the affected organ system
Death-unknown cause (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — specific Adverse Event Terms are unknown because adverse events were only collected with regard to the affected organ system
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — specific Adverse Event Terms are unknown because adverse events were only collected with regard to the affected organ system
Gastrointestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — specific Adverse Event Terms are unknown because adverse events were only collected with regard to the affected organ system
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prequit Combined Nicotine Patch + Gum (N=133) | Prequit Nicotine Patch Only (N=132) | Prequit Nicotine Gum Only (N=131) | No Medication (N=121)
Dizziness (Nervous system disorders) | 12 | 9 | 0 | 0
Headache (Nervous system disorders) | 14 | 15 | 4 | 0
Indigestion (Gastrointestinal disorders) | 15 | 2 | 15 | 0
Insomnia (Nervous system disorders) | 12 | 18 | 3 | 0
Irregular Heartbeat (Cardiac disorders) | 8 | 2 | 3 | 0
Itches or Hives (Skin and subcutaneous tissue disorders) | 6 | 13 | 1 | 0
Mouth Problems (Gastrointestinal disorders) | 5 | 1 | 8 | 0
Nausea (Gastrointestinal disorders) | 18 | 15 | 15 | 0
Skin Rash (Skin and subcutaneous tissue disorders) | 34 | 24 | 0 | 0
VividDreams (Nervous system disorders) | 17 | 26 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes